CLINICAL TRIAL: NCT00906048
Title: A National, Multicenter, Non-comparative Study Evaluating the Efficacy of the Combination of Levofloxacin (500 mg) and Rifampicin (600 or 900 mg Depending on Weight) Administered Once Daily by Oral Route, as Replacement of Empirical Antibiotic Therapy Given Intravenously With a Total Duration of 6 Weeks of the Antibiotic Therapy, in the Treatment of OsteoArticular Prosthetic Infections (OAPI), With a Two-stage Revision of the Prosthesis.
Brief Title: LEVOS - Levofloxacin and Rifampicin Therapy in the Treatment of OsteoArticular Prothethic Infection
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: lack of recruitment
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LEVOF_L_03815; 2008-003284-39(EudraCT)
Record Dates: First submitted 2009-05-20; First posted 2009-05-21 (Estimated); Last update posted 2011-02-07 (Estimated); Status verified 2011-02

CONDITIONS: Infection
MeSH Terms: conditions — Infections | interventions — Levofloxacin

ARMS (1):
- 1 (Experimental): Levofloxacin and Rifampicin
  Interventions: Drug: Levofloxacin (HR355) and Rifampicin Therapy

INTERVENTIONS:
Drug: Levofloxacin (HR355) and Rifampicin Therapy — Film-coated scored tablet measured at 500 mg of levofloxacin and capsule at 300 mg of rifampicin per os once a day
  Weight < 70 kg: 1 tablet of levofloxacin and 2 capsules of rifampicin Weight > 70 kg: 1 tablet of levofloxacin and 3 capsules of rifampicin

SUMMARY:
The primary objective is: to assess the microbiological success of the combination of levofloxacin and rifampicin, administered for 32 to 37 days, as oral replacement therapy of an empirical antibiotic therapy of a maximum of 5 to 10 days given intravenously, in the treatment of OsteoArticular Prosthetic Infections (OAPI), with a two-stage revision of the prosthesis.

The secondary endpoints are:

* To assess the rate of clinical failure 12 months after the reimplantation of the prosthesis.
* To assess the joint mobility function score 12 months after the reimplantation of the prosthesis.
* To assess the safety of the combination of levofloxacin and rifampicin.
* To investigate prognostic factors for success after the end of treatment and at 12 months after the reimplantation of the prosthesis.

ELIGIBILITY:
Inclusion criteria:

* Osteoarticular prosthetic bacterial infection (hip or knee)
* Documented microbiological infection due to Staphylococcus aureus and/or coagulase-negative staphylococci, susceptible to fluoroquinolones and to rifampicin with:

  * For Staphylococcus aureus, a minimum of 2 positive perioperative samples is required.
  * For the coagulase-negative staphylococci, a minimum of 3 positive perioperative samples is required. In the event of combination, there is a minimum of 2 positive perioperative samples for Staphylococcus aureus and a minimum of 3 positive perioperative samples for coagulase-negative staphylococci.
* Two-stage surgical management with: during the first operative stage: removal of the prosthesis, large debridement, implantation or not of a spacer during the second operative stage: implantation of a new cemented prosthesis or not (If possible, without antibiotics as recommended by Sofcot (25), otherwise containing gentamicin).
* Negative urine pregnancy test for females of child-bearing age.
* A barrier contraception method throughout the duration of treatment and for the 4 weeks following the discontinuation of rifampicin for females of child-bearing age.

Exclusion criteria:

* Osteoarticular prosthetic infection at more than one site.
* Osteoarticular prosthetic infection without bacteriological documentation.
* Infection due to staphylococci that are not susceptible to fluoroquinolones or rifampicin.
* Infection not due to staphylococci.
* Absence of surgical management.
* More than 2 surgical repeats due to infection at the infected site.
* Renal impairment with creatinine clearance < 50 ml/min.
* Hepatic impairment.
* Hypersensitivity to levofloxacin, to a product in the quinolone class, to rifamycins or to the excipients of the study products.
* A history of tendinopathy associated with a fluoroquinolone.
* Glucose-6-phosphate dehydrogenase deficiency.
* History of convulsions or epilepsy predisposing factors for the occurrence of convulsions.
* Porphyria.
* Combination use with protease inhibitors or with delavirdine or nevirapine.
* Estrogen-progestin and progestin contraceptives.
* Patient over 65 years of age and who has received corticosteroids.
* Breast-feeding female.
* Pregnant female or female who is likely to become pregnant.
* HIV infection.
* Inflammatory rheumatism.
* Treatment with immunosuppressive agents, cardiovascular, neurological or endocrine disease, or other medically significant disease (cancer, etc.) making the conduct of the protocol or the interpretation of the results of the trial difficult.
* A history of abuse of medicinal products or of alcohol.
* A patient who may receive treatments that are not authorized by the protocol during the trial.
* Treatment with another product undergoing pharmaceutical development during the 4 weeks prior to inclusion in the trial.
* Patient participating in another trial.
* Patient who is allergic to gentamicin, in the event of implantation of a spacer or of cement with gentamicin.
* Mental condition making the patient incapable of understanding the nature, objectives and possible consequences of the trial.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-04; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Microbiological success defined as the percentage of patients with negative peri-operative bacteriological samples and the absence of clinical, biological or radiological signs of infection. | During the reimplantation of the new prosthesis i.e. 15 days to 3 months after the end of treatment

SECONDARY OUTCOMES:
Clinical failure | 12 months after reimplantation of the prosthesis
Joint mobility function score | 12 months after reimplantation of the prosthesis

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Billon, Study Director — sanofi-aventis administrative office
Locations (1):
- Sanofi-Aventis Administrative Office, Paris, France